CLINICAL TRIAL: NCT00433498
Title: A Multicentre Phase III Randomized Double Blind Placebo Controlled Trial of Pravastatin Added to First-Line Standard Chemotherapy in Patients With Small Lung Cancer
Brief Title: Etoposide and Cisplatin or Carboplatin as First-Line Chemotherapy With or Without Pravastatin in Treating Patients With Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000531141; CRUK-LUNGSTAR; EU-20649; ISRCTN56306957; EUDRACT-2005-005821-71; UCL-BRD/05/129; MREC-06-MRE10-28; CTA-20363-0215-001; CTAAC-C1312-A5335; CTAAC-C1312-A12462
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2013-01

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Cisplatin; etoposide phosphate; Pravastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carboplatin/cisplatin and Etoposide with Pravastatin (Experimental)
  Interventions: Drug: carboplatin; Drug: cisplatin; Drug: etoposide phosphate; Drug: pravastatin sodium
- Carboplatin/cisplatin and Etoposide with Placebo (Placebo Comparator)
  Interventions: Drug: carboplatin; Drug: cisplatin; Drug: etoposide phosphate

INTERVENTIONS:
Drug: carboplatin — Should be given according to local practice but suggested doses and schedules are provided in the protocol.
Drug: cisplatin — Should be given according to local practice but suggested doses and schedules are provided in the protocol.
Drug: etoposide phosphate — Day 1: given by IV, days 2 and 3 given by IV or oral. Dose should be given according to local practice but suggested doses and schedules are provided in the protocol.
Drug: pravastatin sodium — 40mg daily oral tablet taken for a maximum of 2 years
  Arms: Carboplatin/cisplatin and Etoposide with Pravastatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as etoposide, cisplatin, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Pravastatin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by making tumor cells more sensitive to chemotherapy. It is not yet known whether etoposide and cisplatin or carboplatin are more effective with or without pravastatin in treating small cell lung cancer.

PURPOSE: This randomized phase III trial is studying etoposide and cisplatin or carboplatin to see how well they work when given as first-line chemotherapy together with pravastatin compared with first-line chemotherapy and a placebo in treating patients with small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the survival of patients with small cell lung cancer treated with etoposide phosphate in combination with cisplatin or carboplatin as first-line chemotherapy with vs without pravastatin.

Secondary

* Compare the progression-free survival of patients treated with these regimens.
* Compare the local progression-free survival (local control) of these patients.
* Compare the response rate in these patients.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to disease stage (limited stage vs extensive stage), ECOG performance status (0 or 1 vs 2 or 3), and participating site. Patients are randomized to 1 of 2 treatment arms.

All patients receive chemotherapy comprising cisplatin IV or carboplatin IV on day 1 and etoposide phosphate IV on days 1-3 or orally twice daily on days 2 and 3. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

* Arm I: Patients receive oral pravastatin daily beginning on day 1 of chemotherapy and continuing for up to 24 months.
* Arm II: Patients receive oral placebo daily beginning on day 1 of chemotherapy and continuing for up to 24 months.

Some patients may undergo blood and urine sample collection at baseline and periodically during and after study treatment. Samples are examined by genetic analysis, metabonomics and proteomics (to detect expression of RAS proteins, phospho-Erk, and other signals downstream of RAS), and cholesterol measurements.

After completion of study treatment, patients are followed every 2 months for 1 year and every 3 months thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

PROJECTED ACCRUAL: A total of 842 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer

  * Limited stage or extensive stage disease
* No mixed cell histology
* No symptomatic brain metastases that require immediate radiotherapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Life expectancy > 8 weeks
* Platelet count > 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count > 1,500/mm^3
* Glomerular filtration rate ≥ 50 mL/min
* Creatine kinase ≤ 5 times upper limit of normal (ULN)
* Liver function tests (ALP, ALT/AST, and bilirubin) < 3 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 1 year after completion of chemotherapy/radiotherapy and for an additional 28 days after completion of pravastatin sodium
* Able to tolerate chemotherapy
* No evidence of significant medical condition or laboratory finding that, in the opinion of the investigator, would preclude study participation
* No family history of hypercholesterolemia
* No history of malignant tumor unless the patient has been without evidence of disease for ≥ 3 years or tumor was a nonmelanoma skin tumor or early cervical cancer

PRIOR CONCURRENT THERAPY:

* More than 12 months since prior statin
* More than 4 weeks since prior fibrates (e.g., bezofibrate, gemfibrozil, or fenofibrate)
* No prior chemotherapy for this cancer
* No prior radiotherapy for this cancer unless to distant metastases (i.e., not within the thorax or thoracic/cervical spine area)
* No concurrent cyclosporine
* Concurrent radiotherapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 846 (Actual)
Dates: Start 2007-01; Primary Completion 2012-01 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Survival | Reported at death.

SECONDARY OUTCOMES:
Progression-free survival | Time until the date of disease progression
Local progression-free survival (local control) | Time until the date of disease progression
Response rate as measured by RECIST criteria after course 3 | Post chemo cycle 3
Toxicity as measured by CTCAE version 3.0 | At every clinic visit or if serious, an SAE form shoudl be submitted

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Seckl, MD, PhD, Study Chair — Charing Cross Hospital
Locations (86):
- United Kingdom (86):
  - William Harvey Hospital, Ashford-Kent, England
  - Stoke Mandeville Hospital, Aylesbury-Buckinghamshire, England
  - North Devon District Hospital, Barnstaple, England
  - Royal United Hospital, Bath, England
  - City Hospital - Birmingham, Birmingham, England
  - Sandwell General Hospital, Birmingham, England
  - Good Hope Hospital, Birmingham, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Bradford Royal Infirmary, Bradford, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Queen's Hospital, Burton-on-Trent, England
  - Addenbrooke's Hospital, Cambridge, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Broomfield Hospital, Chelmsford, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Essex County Hospital, Colchester, England
  - Queen Alexandra Hospital, Cosham, England
  - Darent Valley Hospital, Dartford Kent, England
  - Royal Derby Hospital, Derby, England
  - Dorset County Hospital, Dorchester, England
  - University Hospital of North Durham, Durham, England
  - Princess Alexandra Hospital, Essex, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Gloucestershire Royal Hospital, Gloucester, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Harrogate District Hospital, Harrogate, England
  - Hereford Hospitals, Hereford, England
  - Wycombe General Hospital, High Wycombe, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Castle Hill Hospital, Hull, England
  - Ipswich Hospital, Ipswich, England
  - Airedale General Hospital, Keighley, England
  - Queen Elizabeth Hospital, Kings Lynn, England
  - Cancer Research UK Clinical Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - University College Hospital, London, England
  - Guy's Hospital, London, England
  - Queen Elizabeth Hospital - Woolwich, London, England
  - St. George's Hospital, London, England
  - Charing Cross Hospital, London, England
  - Luton and Dunstable Hospital, Luton, England
  - Maidstone Hospital, Maidstone, England
  - Christie Hospital, Manchester, England
  - Wythenshawe Hospital, Manchester, England
  - Queen Elizabeth The Queen Mother Hospital, Margate, England
  - James Cook University Hospital, Middlesbrough, England
  - Milton Keynes General Hospital, Milton Keynes, England
  - Freeman Hospital, Newcastle upon Tyne, England
  - St. Mary's Hospital, Newport, England
  - Friarage Hospital, North Yorks, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Northampton General Hospital, Nottingham, England
  - Nottingham City Hospital, Nottingham, England
  - King's Mills Hospital, Nottinghamshire, England
  - Princess Royal University Hospital, Orpington, Kent, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Derriford Hospital, Plymouth, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Salisbury District Hospital, Salisbury, England
  - Scarborough General Hospital, Scarborough, England
  - Scunthorpe General Hospital, Scunthorpe, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - South Tyneside District Hospital, South Shields, England
  - Southampton General Hospital, Southampton, England
  - Lister Hospital, Stevenage, England
  - Torbay Hospital, Torquay, England
  - Walsall Manor Hospital, Walsall, England
  - Weston General Hospital, Weston-super-Mare, England
  - New Cross Hospital, Wolverhampton, England
  - Worcestershire Royal Hospital, Worcester, England
  - Worthing Hospital, Worthing, England
  - Yeovil District Hospital, Yeovil, England
  - Cancer Care Centre at York Hospital, York, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Falkirk and District Royal Infirmary, Falkirk, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Llandough Hospital, Cardiff, Wales
  - Nevill Hall Hospital, Gwent, Wales
  - Withybush General Hospital, Haverfordwest, Wales
  - Royal Gwent Hospital, Newport Gwent, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - Singleton Hospital, Swansea, Wales